CLINICAL TRIAL: NCT00852397
Title: A Phase 2, Placebo-Controlled, Randomized, Double-Blinded, Multicenter, Study To Evaluate The Bleeding Profile Of 2.5 Mg And 5.0 Mg BID Apixaban In Combination With Standard Therapy In Patients With Recent (≤7 Days) Acute Coronary Syndrome (ACS)
Brief Title: A Study to Evaluate the Safety of Apixaban in Acute Coronary Syndrome (ACS) Japanese Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B0661004
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Results first posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Apixaban 2.5 mg (Experimental)
  Interventions: Drug: Apixaban
- Apixaban 5.0 mg (Experimental)
  Interventions: Drug: Apixaban
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Apixaban — Apixaban 2.5 mg tablet BID for 24 weeks
  Arms: Apixaban 2.5 mg
Drug: Apixaban — Apixaban 5.0 mg tablet BID for 24 weeks
  Arms: Apixaban 5.0 mg
Other: Placebo — Placebo tablet for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the bleeding safety (the composite endpoint of major and clinically relevant non-major bleeding) of 2 doses of apixaban (2.5 mg BID and 5.0 mg BID) or placebo in combination with standard therapy (aspirin and /or additional antiplatelet therapy) over a 24 week treatment period in selected subjects with recent (≤7 days) acute coronary syndrome.

DETAILED DESCRIPTION:
Due to withdraw of global phase 3 study (APPRAISE-2) for safety issue, B0661004 Data monitoring committee (DMC) also recommended terminating this study. Therefore, Pfizer decided to stop this study.

ELIGIBILITY:
Inclusion Criteria:

* Recent (≤ 7 days) ACS
* Clinically stable, and receiving standard treatment (patients must be treated with aspirin ≤ 100 mg/day, with or without clopidogrel 75 mg/day or ticlopidine 200 mg/day) based on the physician's judgment)

Exclusion Criteria:

* Scheduled/planned cardiac catheterization, PCI, CABG or other invasive procedure planned in the 24 weeks (within treatment period) following randomization
* Persistent severe hypertension, defined as systolic blood pressure of ≥180 mm Hg or diastolic pressure of ≥110 mm Hg
* Active bleeding or at high risk for bleeding (e.g., cirrhosis of the liver, any history of intracranial hemorrhage).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Japan (18):
  - Pfizer Investigational Site, Kasuga, Fukuoka
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Gifu, Gifu
  - Pfizer Investigational Site, Hiroshima, Hiroshima
  - Pfizer Investigational Site, Kure, Hiroshima
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Kumamoto, Kumamoto
  - Pfizer Investigational Site, Uji, Kyoto
  - Pfizer Investigational Site, Ikoma, Nara
  - Pfizer Investigational Site, Hirakata, Osaka
  - Pfizer Investigational Site, Kawachi-Nagano, Osaka
  - Pfizer Investigational Site, Matsubara, Osaka
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Yao, Osaka
  - Pfizer Investigational Site, Wako, Saitama
  - Pfizer Investigational Site, Sunto, Shizuoka
  - Pfizer Investigational Site, Minato-Ku, Tokyo
  - Pfizer Investigational Site, Shinagawa, Tokyo

REFERENCES:
- [Derived] Ogawa H, Goto S, Matsuzaki M, Hiro S, Shima D; APPRAISE-J investigators. Randomized, double-blind trial to evaluate the safety of apixaban with antiplatelet therapy after acute coronary syndrome in Japanese patients (APPRAISE-J). Circ J. 2013;77(9):2341-8. doi: 10.1253/circj.cj-13-0209. Epub 2013 Jun 7. PMID 23748920
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0661004&StudyName=A%20study%20to%20evaluate%20the%20safety%20of%20Apixaban%20in%20Acute%20Coronary%20Syndrome%20%28ACS%29%20Japanese%20patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo was administered twice a day in addition to the standard therapy (aspirin with or without clopidogrel or ticlopidine) for 24 weeks.
- Apixaban 2.5 mg BID: Apixaban 2.5 mg was administered twice a day in addition to the standard therapy (aspirin with or without clopidogrel or ticlopidine) for 24 weeks.
- Apixaban 5.0 mg BID: Apixaban 5.0 mg was administered twice a day in addition to the standard therapy (aspirin with or without clopidogrel or ticlopidine) for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Apixaban 2.5 mg BID | Apixaban 5.0 mg BID
Started | 52 | 49 | 50
Treated Participants | 51 | 49 | 49
Completed | 41 | 41 | 36
Not Completed | 11 | 8 | 14
Not completed — Adverse Event | 4 | 6 | 4
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 2
Not completed — Study terminated by sponsor | 2 | 1 | 6
Not completed — Difficulty in study site visit | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo was administered twice a day in addition to the standard therapy (aspirin with or without clopidogrel or ticlopidine) for 24 weeks.
  Number of participants in baseline characteristics means randomized participants.
- Apixaban 2.5 mg BID: 2.5 mg was administered twice a day in addition to the standard therapy (aspirin with or without clopidogrel or ticlopidine) for 24 weeks.
  Number of participants in baseline characteristics means randomized participants.
- Apixaban 5.0 mg BID: Apixaban 5.0 mg was administered twice a day in addition to the standard therapy (aspirin with or without clopidogrel or ticlopidine) for 24 weeks.
  Number of participants in baseline characteristics means randomized participants.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apixaban 2.5 mg BID | Apixaban 5.0 mg BID | Total
Number analyzed (Participants) | 52 | 49 | 50 | 151
Age Continuous [Mean (Standard Deviation); unit: years] | 63.9 (10.1) | 66.0 (9.0) | 64.0 (9.2) | 64.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 4 | 20
  Male | 42 | 43 | 46 | 131

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had Composite of International Society on Thrombosis and Haemostasis (ISTH)-Defined Major and Clinically-relevant Non-major (CRNM) Bleeding Events Occurring During the Treatment Period.
Description: Major bleeding event was acute clinically overt bleeding accompanied by decrease in hemoglobin of 2 g/dL or more over a 24-hour period, transfusion of 2 or more units of packed red blood cells, or bleeding that occurs in critical site (e.g., intracranial). Fatal bleeding was also major bleeding event. CRNM bleeding was acute or sub-acute clinically overt bleeding that did not satisfy the criteria for major bleeding and that led to either hospital admission for bleeding, physician guided medical or surgical treatment for bleeding or a change in antithrombotic therapy.
Time Frame: Week 0 to Week 24
Population: Bleeding endpoint was included in safety evaluations. The safety analysis set was defined as all treated participants (randomized participants who received at least one dose of study drug).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apixaban 2.5 mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 51 | 49 | 49
Percentage of Participants | 2.0 [0.10 to 9.82] | 4.1 [0.73 to 13.34] | 4.1 [0.73 to 13.34]

2. Secondary Outcome: Percentage of Participants Who Had One or More All Bleeding Occurring During the Treatment Period.
Description: All bleeding included major bleeding (including fatal bleeding), clinically-relevant non-major (CRNM) bleeding, and minor bleeding per international society on thrombosis and haemostasis (ISTH) definitions.
Time Frame: Week 0 to Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apixaban 2.5 mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 51 | 49 | 49
Percentage of Participants | 33.3 [20.76 to 47.23] | 38.8 [26.01 to 53.76] | 44.9 [30.83 to 59.77]

3. Secondary Outcome: Percentage of Participants Who Had Major Bleeding Occurring During the Treatment Period Per International Society on Thrombosis and Haemostasis (ISTH) Definitions.
Description: Major bleeding event was defined as an acute clinically overt bleeding accompanied by decrease in hemoglobin of 2 g/dL or more over a 24-hour period, transfusion of 2 or more units of packed red blood cells, or bleeding that occured in critical site (e.g., intracranial). Fatal bleeding was also major bleeding event.
Time Frame: Week 0 to Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apixaban 2.5 mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 51 | 49 | 49
Percentage of Participants | 0 [0.00 to 6.31] | 2.0 [0.10 to 10.24] | 4.1 [0.73 to 13.34]

4. Secondary Outcome: Percentage of Participants Who Had Thrombolysis in Myocardial Infarction (TIMI)-Defined Major Bleeding Occurring During the Treatment Period.
Description: TIMI major bleeding event was difined as an intracranial bleeding or clinically overt bleeding (including bleeding evident on imaging studies) associated with a >= 5 gm/dL fall in hemoglobin or a 15% fall in hematocrit from baseline, accounting for the effect of transfusions (1 unit packed red blood cells = 1 gm/dL hemoglobin = 3% hematocrit).
Time Frame: Week 0 to Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apixaban 2.5 mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 51 | 49 | 49
Percentage of Participants | 0 [0.00 to 6.31] | 2.0 [0.10 to 10.24] | 2.0 [0.10 to 10.24]

5. Secondary Outcome: Percentage of Participants Who Had Composite of All-cause Death, Non-fatal Myocardial Infarction, Unstable Angina and Stroke During 30 Days After Discontinuation of Therapy.
Time Frame: For 30 days after Week 24 or the discontinuation of study drug
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apixaban 2.5 mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 51 | 49 | 49
Percentage of Participants | 0 [0.00 to 6.31] | 0 [0.00 to 6.53] | 2 [0.10 to 10.24]

6. Secondary Outcome: Percentage of Participants Who Had Composite of All-cause Death, Non-fatal Myocardial Infarction (MI), Unstable Angina, and Non-hemorrhagic Stroke Occurring During the Intended Treatment Period.
Description: Intended treatment period for efficacy endpoints was defined as a period starting on the day of randomization and ending at the later date of either 2-days after the last dose of study drug or Day 168/Week 24 after randomization day (or the study termination date [19 November 2010, Japan time]).
Time Frame: From the day of randomization to the later date of either 2-days after the last dose of study drug or Day 168/Week 24 after randomization day (or the study termination date [19 November 2010, Japan time])
Population: The efficacy analysis set was all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apixaban 2.5 mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 52 | 49 | 50
Percentage of Participants | 1.9 [0.10 to 9.63] | 0 [0.00 to 6.53] | 2.0 [0.10 to 10.03]

7. Other Pre Specified Outcome: Percentage of Participants Who Had International Society on Thrombosis and Haemostasis (ISTH)-Defined Individual Bleeding Endpoints (Clinically-relevant Non-major [CRNM] or Minor Bleeding) During the Treatment Period.
Description: ISTH-defined CRNM bleeding was defined as an acute or sub-acute clinically overt bleeding that did not satisfy the criteria for major bleeding and that led to either hospital admission for bleeding, physician guided medical or surgical treatment for bleeding or a change in antithrombotic therapy.
  ISTH defined minor bleeding event was defined as all acute clinically overt bleeding events not meeting the criteria for either major bleeding or CRNM bleeding were classified as minor bleeding.
Time Frame: Week 0 to Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apixaban 2.5 mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 51 | 49 | 49
Percentage of Participants
  ISTH defined CRNM | 2.0 [0.10 to 9.82] | 2.0 [0.10 to 10.24] | 0 [0.00 to 6.53]
  ISTH defined minor bleeding | 31.4 [19.63 to 45.07] | 36.7 [23.64 to 51.64] | 40.8 [27.00 to 55.79]

8. Other Pre Specified Outcome: Percentage of Participants Who Had Thrombolysis in Myocardial Infarction (TIMI) Defined-individual Bleeding Endpoints (Minor or Minimal Bleeding) During the Treatment Period.
Description: TIMI minor bleeding event was defined as a clinically overt bleeding (including bleeding evident on imaging studies) associated with a >= 3 gm/dL fall in hemoglobin or a 9% fall in hematocrit from baseline, accounting for the effect of transfusions (1 unit packed red blood cells = 1 gm/dL hemoglobin = 3% hematocrit).
  TIMI minimal bleeding event was defined as a clinically overt bleeding (including bleeding evident on imaging studies) not meeting criteria for TIMI minor bleeding.
Time Frame: Week 0 to Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apixaban 2.5 mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 51 | 49 | 49
Percentage of Participants
  TIMI defined minor bleeding | 0 [0.00 to 6.31] | 2.0 [0.00 to 6.53] | 2.0 [0.10 to 10.24]
  TIMI defined minimal bleeding | 33.3 [20.76 to 47.23] | 38.8 [26.01 to 53.76] | 40.8 [27.00 to 55.79]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Apixaban 2.5 mg BID | Apixaban 5.0 mg BID
Serious Adverse Events (participants affected / at risk) | 8/51 | 11/49 | 7/49
Other Adverse Events (participants affected / at risk) | 22/51 | 28/49 | 22/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Apixaban 2.5 mg BID (N=49) | Apixaban 5.0 mg BID (N=49)
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 1 | 1
Arteriospasm coronary (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0
Arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 2 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Apixaban 2.5 mg BID (N=49) | Apixaban 5.0 mg BID (N=49)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3
Gingival bleeding (Gastrointestinal disorders) | 0 | 2 | 3
Chest discomfort (General disorders) | 4 | 1 | 4
Nasopharyngitis (Infections and infestations) | 4 | 4 | 8
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 6 | 6 | 4
Blood urine present (Investigations) | 0 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 2
Headache (Nervous system disorders) | 4 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 4 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.